CLINICAL TRIAL: NCT03548051
Title: Phase 1/2 Placebo Controlled, Partially-Blinded Clinical Trial to Assess the Safety and Efficacy of Microbial Restoration by Enema With Banked and Thawed Processed Stool in Individuals With One or More Recurrences of Clostridium Difficile Associated Disease (CDAD)
Brief Title: Safety and Efficacy of FMT in Individuals With One or More Recurrences of Clostridium Difficile Associated Disease (CDAD)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Low enrollment
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 13-0045; HHSN272201300017I
Record Dates: First submitted 2018-05-24; First posted 2018-06-06 (Actual); Results first posted 2022-05-02 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2021-08-18

CONDITIONS: Clostridial Infection; Dysbiosis; Probiotic Therapy
Keywords: Clinical Trial; Clostridium difficile; Clostridium difficle Associated Disease (CDAD); Efficacy; Fecal Microbiota Transplantation (FMT); Microbial Restoration; Partially-Blinded; Placebo; Safety; Stool
MeSH Terms: conditions — Clostridium Infections; Dysbiosis | interventions — Fecal Microbiota Transplantation; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- FMT group (Experimental): 100 grams of thawed processed stool diluted into 250 ml of saline and delivered by retention enema given 1-3 hours after loperamide 4 mg po x 1, n=108
  Interventions: Procedure: Fecal Microbiota Transplantation (FMT)
- Placebo group (Experimental): 250 ml of saline delivered by retention enema given 1-3 hours after loperamide 4 mg po x 1; if no improvement followed by FMT (100 grams of thawed processed stool diluted into 250 ml of saline and delivered by retention enema given 1-3 hours after loperamide 4 mg po x 1) x 2, n=54
  Interventions: Procedure: Fecal Microbiota Transplantation (FMT); Drug: Saline

INTERVENTIONS:
Procedure: Fecal Microbiota Transplantation (FMT) — 100 grams of thawed processed stool diluted into 250 ml of saline and delivered by retention enema
Drug: Saline — 250 ml of saline delivered by retention enema
  Arms: Placebo group

SUMMARY:
Multi-center, randomized, placebo controlled, partially blinded trial comparing the safety and efficacy of fecal microbiota transplantation versus placebo both delivered by rectal enema in subjects 18 years of age or older with recurrent Clostridium difficile Associated Disease (CDAD). 162 male or female subjects will be enrolled in the study. Enrolled subjects will be randomized at each site to receive either FMT by enema or placebo by enema in a 2:1 ratio. Study duration is 3 years, subject participation duration is approximately 1 year. The primary study objectives are: 1) to evaluate the safety of FMT(s) delivered by enema vs. placebo delivered by enema and 2) to determine efficacy of FMT delivered by enema vs. placebo delivered by enema.

DETAILED DESCRIPTION:
This is a multi-center, randomized, placebo controlled, partially blinded trial comparing the safety and efficacy of fecal microbiota transplantation versus placebo both delivered by rectal enema in subjects 18 years of age or older with recurrent Clostridium difficile Associated Disease (CDAD). 162 (108 in the FMT group, 54 in the placebo group) male or female subjects will be enrolled in the study. Subjects must have had treatment for most recent CDAD with at least 10 days of either metronidazole po/IV (500 mg tid), oral vancomycin (at least 125 mg qid), or oral fidaxomicin (200 mg bid) and have no diarrheal symptoms (<3 unformed stools per 24 hour period) off antibiotics during the washout period. Enrolled subjects will be randomized at each site to receive either FMT by enema or placebo by enema in a 2:1 ratio. The study is described as partially blinded because by design subjects are to be blinded only to a certain point. Subjects will be followed for clinical response (efficacy) and safety. The study duration is 3 years, subject participation duration is approximately 1 year. The primary study objectives are: 1) to evaluate the safety of FMT(s) delivered by enema vs. placebo delivered by enema and 2) to determine efficacy of FMT delivered by enema vs. placebo delivered by enema. Secondary objectives: 1) to evaluate the sustained clinical response rate of FMTs delivered by enema vs. placebo delivered by enema, 2) to evaluate the rate of recurrent CDAD, and 3) to evaluate the time to recurrent CDAD.

ELIGIBILITY:
Inclusion Criteria:

1. Providing permission to access the medical record.
2. Male or non-pregnant female 18 years or older at the time of enrollment.
3. Able to provide signed and dated informed consent.
4. = / > 2 episodes of Clostridium difficile Associated Disease (CDAD) in the past 12 months, including the last episode if present at screening*.

   *Defined by = / > 1 confirmed positive CDAD by diagnostic methods and another occurrence substantiated by medical history.
5. Completed treatment course of at least 10 days of oral vancomycin, oral/IV metronidazole, or oral fidaxomicin for the most recent episode prior to enrollment.
6. Controlled diarrheal symptoms (<3 unformed stools per 24 consecutive hour period).
7. Deemed likely to survive for 1 year after enrollment.
8. Women of childbearing potential* in sexual relationships with men must use an acceptable method of contraception** from 30 days prior to enrollment until 4 weeks after completing study treatment.

   *Not sterilized via tubal ligation, bilateral oophorectomy, salpingectomy, hysterectomy, or successful Essure(R) placement (permanent, non-surgical, non-hormonal sterilization) with documented radiological confirmation test at least 90 days after the procedure, and still menstruating or < 1 year of the last menses if menopausal. Also includes females who are postmenopausal < 1 year.

   **Includes, but is not limited to, barrier with additional spermicidal foam or jelly, intrauterine device, hormonal contraception (started at least 30 days prior to study enrollment), intercourse with men who underwent vasectomy.
9. Males must agree to avoid impregnation of women between Day 1 and 28 days following each administration of the study product.
10. Negative urine or serum pregnancy test within 24 hours of enrollment and randomization.
11. Is able to provide blood and fecal specimens.
12. Is able to complete a test of comprehension.

Exclusion Criteria:

1. Previous fecal microbiota transplantation (FMT) within the previous 12 months prior to study enrollment.
2. Any heart, lung, pancreas, or intestinal transplant recipient or any HIV positive transplant recipient.* *not excluded from the trial are subjects who are kidney, liver, or liver/kidney transplant recipients AND are more than 6 months from transplantation AND have not had a rejection episode in the past 6 months AND have been stable on immunosuppressive regimen for the past 6 months (any prescription change that is due to change of health care provider, insurance company, etc., or that is done for financial reasons, will not be considered a deviation of this criterion)
3. Requiring antibiotics in the past 2 weeks prior to receiving the enema for a condition other than CDAD or scheduled to be used in the upcoming 2 weeks.
4. Unable to tolerate enema for any reason.
5. Any GI cancer in the past 6 months or any actively treated malignancy.*,** *Not excluded from the trial are subjects with actively treated basal and squamous cell cancers without any systemic treatment.

   **Subjects with recently treated malignancy (past 2 months) should have an absolute neutrophil count = / > 1000 /µL since treatment. Subjects with leukemia can not be enrolled in the study.
6. Patients with a history of severe anaphylactic food allergy.
7. Patients with decompensated cirrhosis.*

   *Decompensated cirrhosis is defined as cirrhosis with any history of the following: variceal hemorrhage, ascites, spontaneous bacterial peritonitis, hepatocellular carcinoma, hepatorenal syndrome, or hepatopulmonary syndrome.
8. Untreated HIV disease.*

   *If no HIV screening results are available in the medical record from within the last six months, a HIV screening test will be performed during screening.
9. Other severe immunosuppression or immunodeficiency conditions.*

   *not excluded from the trial are, subjects who take daily dose of systemic corticosteroid equivalent to <20mg prednisone for any duration, or = / > 20 mg prednisone for <14 days, or alternate-day corticosteroid therapy at any dose, OR methotrexate < / = 0.4 mg/kg/week, OR azathioprine < / = 3 mg/kg/day, OR 6-mercaptopurine < / = 1.5 mg/kg/day.
10. Severe OR acute disease at the time of enrollment.*

    *Temperature >100.4 degrees Fahrenheit (38.0 degrees Celsius) or heart rate less than 45 bpm or greater than 130 bpm, or systolic blood pressure less than 80 mm Hg or greater than 155 mm Hg, or diastolic blood pressure greater than 100 mm Hg, or at the discretion of the investigator.
11. Major surgery of the GI tract in the past 2 months.
12. Having a non tolerance* to or any component of vancomycin, loperamide or GoLYTELY.

    *tolerance is defined as the absence of immunoglobulin E-mediated allergy (e.g., urticaria, angioedema, bronchospasm, or anaphylaxis) and the absence of severe allergy (e.g., Stevens-Johnson syndrome/toxic epidermal necrolysis).
13. Active* inflammatory bowel disease (IBD) including ulcerative colitis, Crohn's disease, indeterminate colitis or celiac disease.

    *Active IBD is defined as any IBD requiring any steroid use in the past 6 months OR any increase in dose or frequency of medications in the past 6 months (any prescription change that is due to change of health care provider, insurance company, etc., or that is done for financial reasons, will not be considered a deviation of this criterion).
14. Uncontrolled irritable bowel syndrome (IBS)* or any active uncontrolled gastrointestinal disorders or diseases.**

    *Uncontrolled IBS refers to any IBS with diarrhea on average more than once a week for the past 3 months prior to last CDAD episode.

    **GI obstruction, ileus, gastric retention, bowel perforation, toxic colitis or toxic megacolon, persistent infectious gastroenteritis, persistent or chronic diarrhea of unknown etiology, or refractory/severe Clostridium difficile infection (severe CDAD identified as leukocytosis with a white blood cell count greater than 15,000 cells/mL or an increase in the serum creatinine level to 1.5 times the premorbid level), chronic diarrhea of unknown cause for 6 weeks or more.
15. Unable to comply with protocol requirements.
16. Participation in any other clinical drug research trial within 30 days prior to enrollment or for 1 year after enrollment that might interfere with the safety and efficacy assessment.
17. A condition that would jeopardize the safety or rights of the subject, would make it unlikely for the subject to complete the study, or would confound the results of the study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-01-11 (Actual); Primary Completion 2021-01-13 (Actual); Study Completion 2021-01-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Emory Vaccine Center - The Hope Clinic, Decatur, Georgia
  - Duke Human Vaccine Institute - Duke Vaccine and Trials Unit, Durham, North Carolina
  - Vanderbilt University Medical Center - Infectious Diseases, Nashville, Tennessee

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were males and non-pregnant females 18 years of age or older who are diagnosed with recurrent CDAD. They were recruited from the community at large around the clinical sites. The enrollment period occurred between 11JAN2019 and 23JAN2020.
Groups:
- FMPE Group: 100 g of thawed, processed stool diluted into 250 ml of saline and delivered by retention enema given 1-3 hours after administering loperamide 4 mg orally
  A single dose of fecal microbial suspension contains 100 g of stool in 250 mL diluent, comprising 12.5% glycerol and 87.5% sterile normal saline buffer (0.9% NaCl).
- FMPP Group: 250 ml of saline delivered by retention enema given 1-3 hours after administering loperamide 4 mg orally
  The placebo microbiota preparation (FMPP) is formulated with 250 mL sterile Sodium Chloride (0.9%, USP), Glycerol (12.5%, USP), 8-12 drops brown food coloring (AmeriColor 204 or similar) and water.
Period: Overall Study
Arm/Group | FMPE Group | FMPP Group
Started | 6 | 4
Completed | 4 | 3
Not Completed | 2 | 1
Not completed — Death | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FMPE Group | FMPP Group | Total
Number analyzed (Participants) | 6 | 4 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.5 (13.0) | 60.5 (15.1) | 50.3 (15.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 5
  Male | 2 | 3 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 3 | 9
  Unknown or Not Reported | 0 | 1 | 1
BMI [Mean (Standard Deviation); unit: kg/m^2] | 22.92 (5.17) | 26.28 (8.83) | 24.41 (6.76)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a New Onset of Related Chronic Medical Condition After Completing Treatment for Recurrent Clostridium Difficile-Associated Diarrhea (CDAD)
Description: New onset of related chronic medical conditions (NOCMCs) through 365 days after completing treatment for recurrent CDAD were reported. NOCMCs were defined as any new ICD-10 diagnosis that is applied to the participant during the duration of the study, after receipt of the study agent, that is expected to continue for at least 3 months and requires continued health care intervention.
Time Frame: Day 1 through Day 365
Population: The safety analysis population included all subjects who received the study treatment and had at least one post-treatment safety assessment.
Measure: Count of Participants; unit: Participants
Groups:
- FMPE Group: 100 g of thawed, processed stool diluted into 250 ml of saline and delivered by retention enema given 1-3 hours after administering loperamide 4 mg orally.
- FMPP Group: 250 ml of saline delivered by retention enema given 1-3 hours after administering loperamide 4 mg orally.
Arm/Group | FMPE Group | FMPP Group
Number analyzed (Participants) | 6 | 4
Participants | 0 | 0

2. Primary Outcome: Number of Participants With a Serious Adverse Event (SAE) After Completing Treatment for Recurrent Clostridium Difficile-Associated Diarrhea (CDAD)
Description: SAEs included any adverse event or suspected adverse reaction which, in the view of the investigator or sponsor, resulted in any of the following: death, life threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, a congenital anomaly/birth defect, persistent or significant disability or incapacity or substantial disruption of the ability to conduct normal life function.
Time Frame: Day 1 through Day 365
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | FMPE Group | FMPP Group
Number analyzed (Participants) | 6 | 4
Participants | 3 | 2

3. Primary Outcome: Number of Participants With an Adverse Event (AE) After Completing Treatment for Recurrent Clostridium Difficile-Associated Diarrhea (CDAD)
Description: Adverse events were defined as any noxious, pathologic, or unintended change in anatomic, physiologic, or metabolic functions, as indicated by physical signs, symptoms, and/or laboratory changes occurring in any phase of the clinical trial, regardless of their relationship to investigational product.
Time Frame: Day 1 through Day 30
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | FMPE Group | FMPP Group
Number analyzed (Participants) | 6 | 4
Participants | 4 | 0

4. Primary Outcome: Number of Participants With Newly Acquired Transmissible Infectious Diseases Which Are Considered Adverse Events of Special Interest (AESI), After Completing Treatment for Recurrent Clostridium Difficile-Associated Diarrhea (CDAD)
Description: Adverse Events of Special Interest were defined as newly acquired transmissible infectious agents or infectious diseases related to study product and the following agents: HIV type 1 and 2, Hepatitis A, B, C, Treponema pallidum, HTLV-1, -2, Cyclospora, Salmonella, Shigella, Campylobacter, E. coli 0157:H7, Shiga-toxin producing E. coli, Ova and enteric parasites including Isospora, Vancomycin-resistant Enterococcus (VRE), extended spectrum beta-lactamase (ESBL), carbapenemase producing gram-negative rods, methicillinresistant Staphylococcus aureus (MRSA), Helicobacter pylori, Rotavirus, Adenovirus, Norovirus, Vibrio, Giardia lamblia, Cryptosporidium, and Microsporidia.
Time Frame: Day 1 through Day 365
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | FMPE Group | FMPP Group
Number analyzed (Participants) | 6 | 4
Participants | 0 | 0

5. Primary Outcome: Proportion of Participants With Clinical Response (Defined as no Recurrence of Clostridium Difficile-Associated Diarrhea (CDAD))
Description: Clinical response was defined as those subjects who have no recurrence of CDAD through Day 30 after completing treatment for recurrent CDAD. CDAD was defined as bowel movements as determined by >=3 unformed stools (soft or watery) within 24 consecutive hours and a positive PCR test for Clostridium difficile.
Time Frame: Day 1 through Day 30
Population: The Modified Intention-to-Treat (mITT) analysis population included all randomized subjects who received the study treatment and were followed through the Day 30 visit. Subjects who were not able to retain at least 50% of the enema within 1-3 hours, and either refused a second enema, or were not able to retain at least 50% of the second enema within 1-3 hours were excluded from this population.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | FMPE Group | FMPP Group
Number analyzed (Participants) | 5 | 4
proportion of participants | 0.80 [0.38 to 0.96] | 0.75 [0.30 to 0.95]
Statistical Analysis 1: Comparison: FMPE Group vs FMPP Group; The null hypothesis is that there is no difference in proportions between study arms, with a two-sided alternative; Test type: Superiority; p > 0.999, Fisher Exact — No adjustment for multiple comparisons was made. The a priori threshold for statistical significance is 0.05; Difference in Proportions = 0.05, 95% CI 2-sided [-0.58 to 0.65]

6. Secondary Outcome: Number of Recurrences of Clostridium Difficile-Associated Diarrhea (CDAD) After Completing Treatment for Recurrent CDAD
Description: Recurrence was defined as the re-establishment of diarrhea (frequency of passed unformed stools, >=3 unformed stools within 24 consecutive hours) with a positive PCR test for C. difficile.
Time Frame: Day 1 through Day 30
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: recurrence of CDAD
Arm/Group | FMPE Group | FMPP Group
Number analyzed (Participants) | 5 | 4
recurrence of CDAD | 0.2 (0.4) | 0.3 (0.5)

7. Secondary Outcome: Number of Recurrences of Clostridium Difficile-Associated Diarrhea (CDAD) After Completing Treatment for Recurrent CDAD
Description: as for outcome 6
Time Frame: Day 1 through Day 60
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: recurrence of CDAD
Arm/Group | FMPE Group | FMPP Group
Number analyzed (Participants) | 5 | 4
recurrence of CDAD | 0.2 (0.4) | 0.3 (0.5)

8. Secondary Outcome: Proportion of Participants With Sustained Clinical Response
Description: Sustained clinical response is defined as those subjects who responded by Day 30 with no recurrence of CDAD through Day 60 after randomization.
Time Frame: Day 1 through Day 60
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | FMPE Group | FMPP Group
Number analyzed (Participants) | 5 | 4
proportion of participants | 0.80 [0.38 to 0.96] | 0.75 [0.30 to 0.95]
Statistical Analysis 1: Comparison: FMPE Group vs FMPP Group; The null hypothesis is that there is no difference in proportions between study arms, with a two-sided alternative; Test type: Superiority; p > 0.999, Fisher Exact — No adjustment for multiple comparisons was made. The a priori threshold for statistical significance is 0.05; Difference in Proportions = 0.05, 95% CI 2-sided [-0.58 to 0.65]

9. Secondary Outcome: Time to First Clostridium Difficile-Associated Diarrhea (CDAD) Reoccurrence (Using the Date of First Positive PCR Post-enema)
Description: The time (in weeks) until first CDAD recurrence was calculated as time from randomization to the end of the interval of ascertainment. Participants without a recurrence were censored at their last known contact date or their Day 60 visit, whichever occurred first.
Time Frame: Day 1 through Day 60 visit windows reported as Weeks 1 through 8, respectively
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | FMPE Group | FMPP Group
Number analyzed (Participants) | 5 | 4
participants
  Week 1 at Risk | 5 | 4
  Week 1 with CDAD | 0 | 0
  Week 1 Censored | 0 | 0
  Week 2 at Risk | 5 | 4
  Week 2 with CDAD | 1 | 1
  Week 2 Censored | 0 | 0
  Week 3 at Risk: number analyzed (Participants) | 4 | 3
  Week 3 at Risk | 4 | 3
  Week 3 with CDAD: number analyzed (Participants) | 4 | 3
  Week 3 with CDAD | 0 | 0
  Week 3 Censored: number analyzed (Participants) | 4 | 3
  Week 3 Censored | 0 | 0
  Week 4 at Risk: number analyzed (Participants) | 4 | 3
  Week 4 at Risk | 4 | 3
  Week 4 with CDAD: number analyzed (Participants) | 4 | 3
  Week 4 with CDAD | 0 | 0
  Week 4 Censored: number analyzed (Participants) | 4 | 3
  Week 4 Censored | 0 | 0
  Week 5 at Risk: number analyzed (Participants) | 4 | 3
  Week 5 at Risk | 4 | 3
  Week 5 with CDAD: number analyzed (Participants) | 4 | 3
  Week 5 with CDAD | 0 | 0
  Week 5 Censored: number analyzed (Participants) | 4 | 3
  Week 5 Censored | 0 | 0
  Week 6 at Risk: number analyzed (Participants) | 4 | 3
  Week 6 at Risk | 4 | 3
  Week 6 with CDAD: number analyzed (Participants) | 4 | 3
  Week 6 with CDAD | 0 | 0
  Week 6 Censored: number analyzed (Participants) | 4 | 3
  Week 6 Censored | 0 | 0
  Week 7 at Risk: number analyzed (Participants) | 4 | 3
  Week 7 at Risk | 4 | 3
  Week 7 with CDAD: number analyzed (Participants) | 4 | 3
  Week 7 with CDAD | 0 | 0
  Week 7 Censored: number analyzed (Participants) | 4 | 3
  Week 7 Censored | 0 | 1
  Week 8 at Risk: number analyzed (Participants) | 4 | 2
  Week 8 at Risk | 4 | 2
  Week 8 with CDAD: number analyzed (Participants) | 4 | 2
  Week 8 with CDAD | 0 | 0
  Week 8 Censored: number analyzed (Participants) | 4 | 2
  Week 8 Censored | 4 | 2
Statistical Analysis 1: Comparison: FMPE Group vs FMPP Group; A Log-Rank permutation test for small samples was used to test the null hypothesis that there is no difference in the time to first CDAD recurrence between treatment arms; Test type: Superiority; p > 0.999, Log Rank — No adjustment for multiple comparisons was made. The a priori threshold for statistical significance is 0.05

ADVERSE EVENTS:
Time Frame: Solicited AEs were collected through 8 days after each enema. Non-serious AEs and abnormal clinical laboratory tests were collected from treatment initiation through 30 days after completing treatment for recurrent CDAD. SAEs, NOCMCs, AESIs, and new onset metabolic syndrome were collected from treatment initiation through 365 days after completing treatment for recurrent CDAD. All-cause mortality was assessed through 365 days after completing treatment for recurrent CDAD.
Description: Solicited AEs included fever, chills, nausea, diarrhea, vomiting, constipation, abdominal cramps, abdominal Bloating, flatulence, malaise, fatigue and loss of appetite. Clinical laboratory tests included potassium, creatinine, liver function tests (ALT), hemoglobin, WBC, neutrophil count, platelets.
Arm/Group | FMPE Group | FMPP Group
All-Cause Mortality (participants affected / at risk) | 1/6 | 1/4
Serious Adverse Events (participants affected / at risk) | 3/6 | 2/4
Other Adverse Events (participants affected / at risk) | 6/6 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FMPE Group (N=6) | FMPP Group (N=4)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0)
Cerebral Haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (3) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FMPE Group (N=6) | FMPP Group (N=4)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal Distention (Gastrointestinal disorders) | 6 (38) | 3 (4)
Abdominal Pain (Gastrointestinal disorders) | 6 (32) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (15) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 4 (11) | 3 (14)
Flatulence (Gastrointestinal disorders) | 4 (23) | 2 (11)
Nausea (Gastrointestinal disorders) | 3 (5) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Chills (General disorders) | 2 (5) | 1 (1)
Malaise (General disorders) | 4 (22) | 1 (2)
Pyrexia (General disorders) | 1 (4) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 3 (15) | 1 (1)
Diastolic Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Systolic Hypertension (Vascular disorders) | 0 (0) | 1 (4)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0)
Blood pressure Increased (Investigations) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2021-08-24): https://cdn.clinicaltrials.gov/large-docs/51/NCT03548051/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-20): https://cdn.clinicaltrials.gov/large-docs/51/NCT03548051/SAP_001.pdf